CLINICAL TRIAL: NCT03530033
Title: Lidocaine Reduces Muscle Tremor Caused by Electric Energy Devices, Which is Beneficial for Intraoperative Recurrent Laryngeal Nerve Monitoring During Endoscopic Thyroid Lateral Neck Dissection
Brief Title: Lidocaine Reduces Muscle Tremor is Beneficial for Intraoperative Recurrent Laryngeal Nerve Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bo Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Bo Wang,MD, clinical Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BND IONM Lidocaine
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Thyroid Cancer; Neck Cancer; Recurrent Laryngeal Nerve Injuries; Accessory Nerve Injuries; EMG: Repetitive Nerve Stimulation Abnormality
MeSH Terms: conditions — Thyroid Neoplasms; Head and Neck Neoplasms; Recurrent Laryngeal Nerve Injuries; Accessory Nerve Injuries | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional surgery group (No Intervention): Induction of anesthesia according to conventional neuromuscular blockade dose, no neuromuscular blockade drug maintenance during lateral neck dissection.
- Lidocaine group (Experimental): Anesthesia induction was performed according to conventional nerve monitoring neuromuscular blockade doses and lateral neck dissection was performed. When local muscle tremors occur, lidocaine is injected locally to eliminate muscle tremors.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Local injection of lidocaine reduces muscle tremor
  Arms: Lidocaine group

SUMMARY:
In recent years, the application of intraoperative recurrent laryngeal nerve monitoring in thyroid surgery has greatly reduced the complications of recurrent laryngeal nerve injury. The use of intraoperative neurological monitoring requires the reduction of the dose of neuromuscular blockade, which often leads to muscle tremors during the application of electrical energy, which affects the fine separation around the muscles. This study explored the effect of local application of lidocaine on reducing muscle tremor during surgery and its optimal dose.

DETAILED DESCRIPTION:
According to the random number method, eligible patients were randomly divided into 2 groups. Group A was the conventional surgery group, and Group B was the lidocaine group. The operative time for the separation of the sternocleidomastoid muscle from the two groups of patients was analyzed, as well as the length of time for the search for the accessory nerve and the effect of intraoperative nerve monitoring on the EMG signal.

ELIGIBILITY:
Inclusion Criteria:

* Thyroid papillary carcinoma
* Lateral cervical lymph node metastasis
* The diameter of the metastatic lymph nodes is less than 3cm
* Without internal jugular vein invasion

Exclusion Criteria:

* Lidocaine allergy sufferers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
dose of muscle relaxant drugs | At the end of surgery
  dose of muscle relaxant drugs
dose of lidocaine | At the end of surgery
  dose of lidocaine
Number of nerve signal loss cases | At the end of surgery
  Number of nerve signal loss cases
Anatomical time of accessory nerve | At the end of surgery
  Anatomical time of accessory nerve
The satisfaction of sternocleidomastoid muscle separation | At the end of surgery
  The visual score was 5 points for the most satisfaction and 0 points for the most dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China